CLINICAL TRIAL: NCT00901927
Title: A Phase II Study of Bendamustine, Mitoxantrone, and Rituximab (BMR) for Patients With Untreated High Risk Follicular Lymphoma
Brief Title: Bendamustine, Mitoxantrone, and Rituximab (BMR) for Patients With Untreated High Risk Follicular Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was closed early due to toxicity
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Cephalon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0204; NCI-2012-01629 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-05-12; First posted 2009-05-14 (Estimated); Results first posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Follicular Lymphoma
Keywords: Lymphoma; Non-Hodgkin's Lymphoma; Untreated High Risk Follicular Lymphoma; Bendamustine hydrochloride; Bendamustine HCI; Bendamustine; CEP-18083; SDX-105; Treanda; Mitoxantrone; Novantrone; Rituximab; Rituxan
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma; Lymphoma, Non-Hodgkin | interventions — Bendamustine Hydrochloride; Mitoxantrone; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bendamustine + Mitoxantrone + Rituximab (Experimental): Bendamustine starting dose 90 mg/m^2 intravenously (IV) over 30-60 minutes on Days 1 and 2 of each 8-day cycle. Mitoxantrone 10 mg/m^2 IV over 15 minutes on Day 2 of each cycle. Rituximab 375 mg/m^2 IV over several hours on Day 1 of each cycle.
  Interventions: Drug: Bendamustine; Drug: Mitoxantrone; Drug: Rituximab

INTERVENTIONS:
Drug: Bendamustine — Starting dose 90 mg/m^2 by vein over 30-60 minutes on Days 1 and 2 of each cycle.
  Other Names: Bendamustine Hydrochloride; Bendamustine HCI; CEP-18083; SDX-105; Treanda
Drug: Mitoxantrone — 10 mg/m^2 by vein over 15 minutes on Day 2 of each cycle.
  Other Names: Novantrone
Drug: Rituximab — 375 mg/m^2 by vein over several hours on Day 1 of each cycle.
  Other Names: Rituxan

SUMMARY:
The goal of this clinical research study is to learn if the combination of bendamustine hydrochloride, mitoxantrone, and rituximab can help to control follicular lymphoma.

The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Bendamustine is designed to damage and destroy the DNA (genetic material) of cancer cells.

Mitoxantrone is designed to stop cancer cells from making DNA, which may stop the cells from making more cells.

Rituximab is designed to attach to lymphoma cells, which may cause them to die.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive the study drugs in 28-day "cycles."

On Days 1 and 2 of each cycle, you will receive bendamustine through a needle in a vein over 30-60 minutes.

On Day 1 of each cycle, you will receive rituximab by vein over several hours, depending on how well you tolerate it. Usually, the first dose of rituximab is given over 6-8 hours. If you tolerate the first dose well, you will receive the next doses over 4 hours.

On Day 2 of each cycle, you will receive mitoxantrone by vein over 15 minutes.

Study Visits:

At every study visit (Days 1, 8, 15, and 22 of each cycle), your vital signs will be measured. You will be asked if you have experienced any side effects and to list any drugs you may be taking. The measurement of vital signs on Days 8, 15, and 22 of each cycle may be done by your personal doctor, and the results can be sent in to the study staff.

On Day 1 of each cycle, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your weight.
* Blood (about 1-2 teaspoons) will be drawn for routine tests.
* You will have a performance status evaluation.

On Days 8, 15, and 22 of each cycles, blood (about 1 teaspoon) will be drawn for routine tests. These tests may be performed by your personal doctor, and the results can be sent in to the study staff.

At the end of Cycle 3, you will have a positron emission tomography (PET) scan and/or CT scan to check the status of the disease.

If your bone marrow showed lymphoma at the beginning of the study, you will have an additional bone marrow aspiration and biopsy if the disease goes away while you are on study. This will be to check the status of the disease.

If at any time the doctor thinks it is necessary, you will have extra blood and urine collected for routine tests.

Length of Study Participation:

You may receive up to 6 cycles (about 6 months) of study treatment. If the disease gets worse or intolerable side effects occur, you will be taken off study treatment early.

End-of-Study Visit:

At 30-40 days after your last dose of study drugs, you will have an end-of-study visit. At this visit, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs and weight.
* You will have a performance status evaluation.
* Blood (about 1-2 teaspoons) will be drawn for routine tests.
* You will have CT and PET scans to check the status of the disease.
* You will be asked if you have experienced any side effects and to list any drugs you may be taking.

Long-Term Follow-Up:

Every 3 months for 2 years after your study treatment ends, you will have follow-up visits. If after 2 years your body shows no signs of cancer, you will have follow-up visits every 6 months after that. These follow-up tests are considered routine care.

The following tests and procedures will be performed at these visits:

* You will have a performance status evaluation.
* Blood (about 1-2 teaspoons) will be drawn for routine tests.
* You will be asked how you are doing and whether you are receiving any new treatments for the disease.
* You will have CT and PET scans to check the status of the disease.
* The study doctor will check the results of any other scans and tests you may have for routine care. The study doctor will also check the results of physical exams you may have.

This is an investigational study. All 3 study drugs are commercially available. Rituximab is FDA approved to treat follicular lymphoma. Mitoxantrone is FDA approved for use in combination for certain types of leukemia. Bendamustine is FDA approved to treat chronic lymphocytic leukemia.

The combination of rituximab, mitoxantrone, and bendamustine is not FDA approved to treat follicular lymphoma. At this time, it is only being used in research.

Up to 37 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years at the time of signing the informed consent form.
2. Able to adhere to the study visit schedule and other protocol requirements.
3. Untreated grade 1, 2, or 3a follicular non-Hodgkin's lymphoma.
4. At least one measurable lesion according to the International Working Group Criteria for Response, of greater that 1.5cm.
5. Eastern Cooperative Oncology Group (ECOG) performance status of < 2 at study entry.
6. Laboratory test results within these ranges: Absolute neutrophil count >/=1.5 x 10^9/L; Platelet count >/=100 x 10^9/L; Serum creatinine </= 2.0 mg/dL; Total bilirubin </= 1.5 mg/dL; AST (SGOT) and ALT (SGPT) </= 2 x upper limit of normal (ULN) or </= 5 x ULN if hepatic metastases are present.
7. Disease free of prior malignancies for at least 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix or breast.
8. Have a high risk FLIPI score, as defined by a FLIPI score >/= 3.
9. Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 milli-International unit (mIU)/mL within 10 to 14 days prior to study entry.
10. An ejection fraction of >/= 50% as documented by a cardiac function study.

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
2. Pregnant or breast feeding females.
3. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
4. Use of any prior chemotherapy for follicular lymphoma.
5. Known hypersensitivity to Bendamustine, mitoxantrone, or mannitol.
6. A history of congestive heart failure.
7. Any prior use of bendamustine or mitoxantrone.
8. Concurrent use of other anti-cancer agents or experimental treatments.
9. Known positive for HIV or infectious hepatitis type B or C.
10. Creatinine clearance less than 40 ml/min.
11. A known history of hepatic insufficiency (patients with a history of fulminate hepatic failure, hepatic encephalopathy, cirrhosis, and autoimmune hepatitis).
12. Any history of grade 3b follicular lymphoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Fowler, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: May 12, 2009 to June 30, 2011. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Groups:
- Bendamustine + Mitoxantrone + Rituximab: Bendamustine, Mitoxantrone, and Rituximab, 6, 28 day cycles
Period: Overall Study
Arm/Group | Bendamustine + Mitoxantrone + Rituximab
Started | 14
Completed | 8
Not Completed | 6
Not completed — Lack of Efficacy | 1
Not completed — Protocol Violation | 3
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Bendamustine + Mitoxantrone + Rituximab
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 4
Age, Continuous [Median (Full Range); unit: years] | 69.5 [50 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate of the Combination of BMR (Bendamustine + Mitoxantrone + Rituximab)
Description: To evaluate the complete response rate of the combination of BMR in previously untreated follicular non-Hodgkin's lymphoma. CR defined by International Working Group Criteria for Response for Non-Hodgkin's Lymphoma as complete disappearance of all detectable clinical evidence of disease and disease-related symptoms.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Bendamustine + Mitoxantrone + Rituximab
Number analyzed (Participants) | 8
participants | 3

2. Secondary Outcome: Participants With Adverse Events
Description: To evaluate the toxicity and safety of BMR in participants with untreated follicular lymphoma.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bendamustine + Mitoxantrone + Rituximab
Number analyzed (Participants) | 8
Participants | 3

3. Secondary Outcome: Time to Progression (TTP) for Participants Treated With BMR (Bendamustine, Mitoxantrone, and Rituximab)
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 5 months
Measure: Median (Full Range); unit: months
Arm/Group | Bendamustine + Mitoxantrone + Rituximab
Number analyzed (Participants) | 8
months | 5 [1 to 9]

ADVERSE EVENTS:
Time Frame: Adverse event collection through each 28 day cycle, up to 6 cycles or 180 days.
Arm/Group | Bendamustine + Mitoxantrone + Rituximab
Serious Adverse Events (participants affected / at risk) | 8/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bendamustine + Mitoxantrone + Rituximab (N=8)
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Fatigue (General disorders) | 1
Hgb Decreased (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 8
Lymphopenia (Blood and lymphatic system disorders) | 1
ANC Decrease (Blood and lymphatic system disorders) | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bendamustine + Mitoxantrone + Rituximab (N=8)
Anxiety (Nervous system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cecal infection (Gastrointestinal disorders) | 1
Chills (General disorders) | 2
Conduction disorder (Cardiac disorders) | 1
Constipation (Gastrointestinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 4
Dry eye syndrome (Eye disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Edema limbs (Musculoskeletal and connective tissue disorders) | 1
Eye pain (Eye disorders) | 1
Fatigue (General disorders) | 6
Fracture (Musculoskeletal and connective tissue disorders) | 1
Glucose intolerance (Endocrine disorders) | 1
Growth and Development (Other) (General disorders) | 1
Hemoglobin decreased (Blood and lymphatic system disorders) | 2
Hypersensitivity (Skin and subcutaneous tissue disorders) | 1
Infection (Other) (Infections and infestations) | 1
Injection site reaction (Skin and subcutaneous tissue disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 1
Localized edema (General disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Memory impairment (Nervous system disorders) | 2
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 8
Neuralgia (Nervous system disorders) | 1
Neutrophil count decreased (Blood and lymphatic system disorders) | 1
Peripheral motor neuropathy (Musculoskeletal and connective tissue disorders) | 1
Petechiae (Blood and lymphatic system disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Serum magnesium decreased (Metabolism and nutrition disorders) | 1
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1
Trismus (Musculoskeletal and connective tissue disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Vaginal infection (Infections and infestations) | 1
Vision blurred (Eye disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Watering eyes (Eye disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes